CLINICAL TRIAL: NCT06856980
Title: Comparative Study Between Syndesmotic Screw and Suture Button in Ankle Syndesmotic Diastasis
Brief Title: Syndesmotic Screw Vs Suture Button in Ankle Syndesmotic Diastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, El-Sayed Sherif Soliman El-Gamasy, Resident of Orthopedic Surgery, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264MS76/6/23
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Syndesmotic Screw; Suture Button; Fixation; Ankle Syndesmotic Diastasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture button fixation (Experimental): Patients undergoing suture button fixation of syndesmosis injury
  Interventions: Procedure: Suture button fixation
- Syndesmotic screw fixation (Experimental): Patients undergoing syndesmotic screw fixation of syndesmosis injury
  Interventions: Procedure: Syndesmotic screw fixation

INTERVENTIONS:
Procedure: Suture button fixation — Patients undergoing suture button fixation of syndesmosis injury.
  Other Names: Group A
  Arms: Suture button fixation
Procedure: Syndesmotic screw fixation — Patients undergoing syndesmotic screw fixation of syndesmosis injury.
  Other Names: Group B
  Arms: Syndesmotic screw fixation

SUMMARY:
The aim of this study is to compare suture-button versus syndesmotic screw in the treatment of distal tibiofibular syndesmotic injury.

DETAILED DESCRIPTION:
The term syndesmotic injury is used to describe a lesion of the ligaments that connect the distal fibula and the tibial notch surrounded on both sides by the anterior and posterior tibial tubercles, with or without an associated injury of the deltoid ligament.

Accuracy and maintenance of syndesmosis reduction are considered the key elements in the treatment of ankle fractures. Screw fixation is considered the gold standard treatment for an unstable syndesmosis injury.

Button and suture construction with a medial-lateral metallic button and suture system offers an alternative method for repairing the distal tibio-fibular joint. Suture-button design has been shown to maintain the reduction, facilitating physiologic stability of the ankle mortise. This may allow early physiological motion, leading to earlier ligament healing and potentially earlier loading, which may produce better clinical results. However, this system is more expensive than the screw method and it may gradually relax under weightbearing conditions. Therefore, whether this device is a suitable alternative, and how many devices are needed for adequate stability are not yet known.

ELIGIBILITY:
Inclusion Criteria:

- Unstable unilateral syndesmotic injuries that was considered by the attending staff surgeon to require surgical fixation, including:

* Age : 18 - 60 years old.
* Closed or grade I open fractures are included.
* Isolated syndesmotic injury.
* associated lateral malleolus fracture with talar shift.
* Associated with Bimalleolar fractures.
* Associated with Trimalleolar fractures that did not require posterior fragment fixation (typically <25% of articular surface).

Exclusion Criteria:

- Exclusion criteria include patient and injury specific factors.

Patient-related exclusion factors included:

* Skeletal immaturity.
* Previous ipsilateral ankle surgery.
* Non-ambulatory status before injury.
* Inability to comply with postoperative protocol (i.e., advanced dementia).
* Medical unfit patients for surgery.
* Uncontrolled diabetes mellitus with charcot joint or peripheral neuropathy.
* Polytrauma patients.

Injury-related exclusion factors included:

* Grade II or III open fractures
* Tibial plafond fractures
* Posterior malleolar fractures requiring fixation (typically >25% articular surface involved).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The American Orthopaedic Foot and Ankle Society (AOFAS) | 12 months postoperatively
  As an interpretation of the American Orthopaedic Foot and Ankle Society (AOFAS) score, excellent results with score between (95-100). Good results between (75-94). Fair results between (51-74). Poor results between (0-50).

SECONDARY OUTCOMES:
Degree of pain | 12 months postoperatively
  Degree of pain was assessed using an interpretation of visual analogue scale (VAS) score, No pain with score 0, mild pain with score between (1-3), moderate pain with score between (4-7) and severe pain with score between (8-10). VAS was assessed at 6 weeks, 6 months and 12 months postoperatively.
Ankle Range of motion (ROM) | 12 months Postoperatively
  Motion of the ankle occurs primarily in the sagittal plane, with plantar- and dorsiflexion occurring predominantly at the tibiotalar joint. Overall Ankle range of motion (ROM) in the sagittal plane of between 65 and 75°, moving from 10 to 20° of dorsiflexion through to 40-55° of plantarflexion.
  Sagittal motion (flexion plus extension) Normal or mild restriction (30° or more) : 8 Moderate restriction (15°-29°) : 4 Severe restriction (less than 15°) : 0

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.